CLINICAL TRIAL: NCT01219361
Title: Evaluation of Donated Human Embryos for Study of Normal and Abnormal Differentiation and Development Following in Vitro Fertilization.
Brief Title: Evaluation of Donated Human Embryos Following in Vitro Fertilization
Status: Enrolling by invitation | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-05
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Validation of Laboratory Techniques; Validation of Laboratory Methods; Assessment of Laboratory Staff Proficiency
Keywords: Donated embryos

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Donated embryos
Oversight: Data Monitoring Committee: No

SUMMARY:
Couples who have created excess embryos while undergoing IVF procedures, and who do not wish to transfer those embryos or donate them to another couple may donate the extra embryos to research. The embryos are then used to develop improved laboratory techniques and conditions as well as testing the proficiency of laboratory staff.

DETAILED DESCRIPTION:
Undergoing IVF treatment often results in the production of more embryos than can safely be transferred at one time. These extra embryos are often cryopreserved for future use. In the event that a couple decides that they do not want to proceed with using cryopreserved embryos, these embryos can be discarded, donated to another couple, or donated to research.

Embryos that are donated to research are used to identify a group of parameters that have significant predictive value for assisted reproductive technology outcomes. We hope to develop future laboratory techniques as we gain a better knowledge of gamete development, fertilization and implantation. We will test, standardize and implement better methods for freezing embryos prior to employing these techniques in a clinical setting. We hope to develop new methods to optimize the determination of genes and chromosomes in embryos. We will test the proficiency of laboratory staff on techniques and/or procedures done in the IVF laboratory. This study WILL NOT:create embryos for research, transfer embryos to an individual, develop cell lines or clones.

ELIGIBILITY:
Inclusion Criteria:

none

Exclusion Criteria:

none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients will cryopreserved embryos who do not want to discard them or donate them to another couple
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2005-07; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Freezing methods for embryos | duration of the study
  To test, standardize and implement better methods for the freezing of embryos prior to these techniques being implemented in the clinical setting.

SECONDARY OUTCOMES:
Development of New Methods | duration of the study
  The development of new methods to optimize the determination of genes and chromosomes in embryos

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Molinaro, MD, MSCE, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Basking Ridge, New Jersey, United States